CLINICAL TRIAL: NCT05908201
Title: Effects of 6-weeks of Early Time Restricted Eating on Muscle Performance in Resistance Trained Individuals
Brief Title: Effects of Early Time Restricted Eating on Muscle Performance in Resistance Trained Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Mississippi, Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-030
Record Dates: First submitted 2023-03-21; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Time Restricted Eating
Keywords: Intermittent fasting; Time restricted eating
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early time-restricted eating (Experimental): The Early Time Restricted Eating (eTRE) group will be asked to consume calorie containing food or drinks only between 9am to 5pm, daily. At other times they are to avoid consuming any calorie containing food or drinks.
  Interventions: Behavioral: early time restricted eating
- Control (No Intervention): The Control group will follow their usual eating routine.

INTERVENTIONS:
Behavioral: early time restricted eating — The intervention group will eat in a prescribed daily feeding window (9am-5pm) and follow their normal exercise and resistance training routines. We will allow up till +/-1 hour for the eating window start and end times while aiming for an 8 hour eating window.
  Arms: early time-restricted eating

SUMMARY:
A randomized controlled trial to determine the effectiveness of early time-restricted eating on muscle performance and body composition in active, resistance trained adults. Two parallel groups will be randomly assigned to either the early time-restricted eating or a control group. All participants will be asked to maintain their usual exercise routines during the 6 week intervention period. Muscle strength and endurance are the primary outcomes. Body composition (body weight, fat mass, fat-free mass and percent body fat), hunger and satiety ratings, sleep quality, energy intake, diet quality, macronutrient composition and adherence are secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 - 50 years
* Performing resistance training at least twice per week (for ≥1 yr)
* BMI ≥ 18.5

Exclusion Criteria:

* Currently sedentary or not engaged in resistance training.
* Major surgeries in muscles/joints during the past 3 months
* BMI < 18.5
* Ineligible to engage in physical activity according to 2022 Physical Activity Readiness Questionnaire for everyone (PAR-Q+)
* Take anabolic steroids or on hormone replacement therapy.
* Current smoker.
* Following restrictive diets (Vegan, vegetarian, intermittent fasting, Paleo, calorie restriction, keto/ low carbohydrate diet or any other restrictive diets)
* Active cancer or cancer requiring treatment in the past 2 years (except non-melanoma skin cancer).
* Musculoskeletal disorders
* Diagnosed with cardiovascular disease including myocardial infarction, heart surgery, heart failure and had a heart transplant.
* Have pacemaker or metal implants
* Diagnosed diabetes (type 1 or 2).
* Diagnosed hypertension or high blood pressure (>130/90).
* Diagnosed eating disorder or score ≥ 20 on Eating Attitudes Test -26 (EAT26) survey
* Missing limbs/ have prosthetics
* Had surgery in joints/muscle in the past year.
* Received medical advise against exercising due to medical reasons.
* On medication for conditions related to the thyroid gland
* Unwilling to commit for a 7-week study
* Likely to move away from participating clinic before trial completed
* Unable or unwilling to give informed consent
* Another household member is a participant or staff member in the trial
* Unwilling to accept treatment assignment by randomization
* Current or anticipated participation in another intervention research project that would interfere with the intervention offered in the trial
* Pregnant or < 6 months since giving birth.
* Any other condition which, in opinion of investigators, that would adversely affect conduct of the trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Muscular strength | 6-weeks
  Pre and post intervention testing of muscular strength using one-rep max
Muscular endurance | 6-weeks
  Pre and post intervention testing of muscular endurance using barbell bench press and squat.

SECONDARY OUTCOMES:
Body weight (kg) | 6-weeks
  Pre and post intervention measures of body weight.
Hunger and satiety | 6-weeks
  Pre and post intervention subjective measure of hunger and satiety with the use of a Hunger and Satiety Visual Analog Scale (minimum value zero, maximum value 10). Higher the score, the more hungry/ less satiated one is.
Sleep quality | 6-weeks
  Pre and post intervention measure of subjective sleep quality by use of Pittsburgh Sleep Quality Scale. (each question can be scored from 0-3, then an aggregate score of the whole survey can range from 0-21; The higher the score the worst the sleep quality).
Total calorie intake | 6-weeks
  Pre and post intervention measurements of calorie intake based on 24-hour food recall survey using the Automated Self-Administered 24-hour (ASA24) software.
Diet Quality | 6-weeks
  Pre and post intervention measurements of diet quality based on 24-hour food recall survey using the ASA24 software and Healthy Eating Index.
Diet macronutrient composition | 6-weeks
  Pre and post intervention measurements of macronutrients based on 24-hour food recall survey using the ASA24 software.
Adherence | 6-weeks
  Percent of days during the 6-week trial when eTRE was adhered to as recommended. This will be recorded by the participants daily throughout the entire study.
Fat mass | 6-weeks
  Pre and post intervention measurements of body fat mass (kg).
Fat-free mass | 6-weeks
  pre and post intervention measurements of body fat-free mass (kg).
Body fat percentage | 6-weeks
  Pre and post intervention measurements of body fat percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition and Hospitality Management, University of Mississippi, University, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share the de-identified participant data used in the published manuscript/s by depositing these data in the Open Science Framework (OSF) repository. The data shared will include the sociodemographic data and the outcomes published in the manuscripts. The protocol and statistical analysis plan will be shared as supplementary material through the journal where the study if published, if allowed.
Supporting Information: Study Protocol, SAP
Time Frame: We agree to deposit outcome data into the OSF repository as soon as possible but no later than within two years after the last publication.